CLINICAL TRIAL: NCT00582907
Title: Phase 2 Study of IL-1 Trap (Rilonacept) for Treatment of Familial Mediterranean Fever (FMF)
Brief Title: Rilonacept for Treatment of Familial Mediterranean Fever (FMF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Philip Hashkes, Study Director, Shaare Zedek Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01FD003435-01 (FDA); FDA 1RO1FD003435-01; NCT00767143 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Familial Mediterranean Fever
Keywords: FMF; IL1 Trap (Rilonacept); Periodic fever syndromes; Autoinflammatory syndromes; Familial Mediterranean Fever; colchicine
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Treatment Arm A: Rilonacept (IL-1 Trap) at a dose of 2.2 mg/kg/wk (max 160 mg)given by subcutaneous injection for 3 months plus colchicine at a stable dose for those subjects already taking colchicine, or without colchicine for those intolerant or non-compliant with colchicine. Since the colchicine dose is stable throughout the study for each subject, at the prestudy dose, colchicine was not considered an intervention
  Interventions: Drug: Rilonacept
- 2 (Placebo Comparator): Treatment Arm B: Placebo given by subcutaneous injection weekly with or without colchicine for 3 months. Since the colchicine dose is stable throughout the study for each subject, at the prestudy dose, colchicine was not considered an intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept — 2.2 mg/kg/wk by subcutaneous injection, for 3 months
  Other Names: Arcalyst, IL-1 Trap
  Arms: 1
Drug: Placebo — placebo by subcutaneous injection weekly for 3 months
  Arms: 2

SUMMARY:
Familial Mediterranean fever (FMF) is a genetic disease resulting in recurrent attacks of fever, abdominal pain, chest pain, arthritis and rash. There are 5-15% of patients who continue to have FMF attacks despite treatment with colchicine or who cannot tolerate colchicine. Currently there are no alternatives to colchicine. Pyrin, the protein that has a defect in FMF has an important role in the regulation of a molecule called interleukin (IL)-1 beta production and activity. This molecule is very important in the process of inflammation in FMF.

Therefore we propose to use IL-1 Trap (Rilonacept), a medication that binds and neutralizes IL-1.

We will enroll in this study 17 subjects from the age of 4 years, including adults with active FMF despite colchicine therapy. Subjects will receive in random order two 3-month courses of Rilonacept at 2.2 mg/kg (maximum 160 mg) by weekly subcutaneous injection and two 3-month courses of placebo injection. If patients have at least two FMF attacks during a treatment course they will be able to get if they choose the other treatment until the end of that treatment course. Our hypothesis is that Rilonacept will decrease the number of acute FMF attacks and will be safe to use. This study may confirm the importance of IL-1 in the cause of FMF.

Funding source - FDA Office of Orphan Products Development

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is an autosomal recessive autoinflammatory genetic disorder resulting in recurrent attacks of fever, serositis, arthritis and rash. Late complications of untreated FMF include the development of renal amyloidosis. FMF is a rare orphan disease in the United States. Treatment with colchicine is effective in reducing the frequency of episodes in most patients and the development of amyloidosis in nearly all patients. However, there are still 5-15% of patients who continue to have acute FMF attacks despite colchicine therapy or are intolerant of colchicine, usually from gastrointestinal adverse effects. Currently there are no effective alternatives to colchicine. Pyrin, the mutated protein in FMF has an important role in the regulation of IL-1 beta production and activity. Mutations in pyrin result in increased IL-1 beta levels in mice and humans. IL-1 beta is an important pro-inflammatory cytokine. Thus, we hypothesize that inhibition of IL-1 will decrease acute attacks in patients with FMF. We propose to use IL-1 Trap (Rilonacept), a fusion protein consisting of human IL-1 cytokine receptor extracellular domains and the FC portion of human IgG1 that binds and neutralizes IL-1.

We will enroll 17 subjects from the age of 4 years, including adults, from multiple centers in the United States with active FMF (at least 1 attack per month) despite receiving at least 1.2-1.5 mg/d of colchicine (dose dependent on age) or are intolerant of colchicine. Subjects will be diagnosed by clinical criteria with at least one heterozygote mutation of the MEFV (pyrin) gene. After screening subjects will be monitored for a month to observe for acute FMF attacks or if they did not develop an attack in that month until they develop two attacks. We will then use a single-subject alternating treatments design with subjects receiving in random order two 3-month courses of Rilonacept at 2.2 mg/kg (max 160 mg) by weekly SC injection and two 3-month courses of comparable volume placebo. Subjects will continue the usual colchicine dose they were on when they started the study. Subjects with 2 acute FMF attacks during a treatment course will be able to crossover to the other treatment arm until the end of that treatment course. There will be 10 study visits: 1. Screening. 2. Treatment baseline after one month or after subjects have developed FMF attacks as described above. After 1 month of each treatment course and at the end of each treatment course (overall 8 visits). At each visit subjects will return completed diary forms, used and unused drug, queried on adverse effects, undergo a physical examination and laboratory tests obtained for inflammation, safety and in some visits for translational studies. Subjects will also fill out quality of life questionnaires and give an overall estimation of the disease activity. Results will be analyzed by traditional frequency statistics (using an intent to treat analysis) and by Bayesian hierarchical modeling. Our primary aim is to assess the efficacy of Rilonacept in decreasing the number of acute FMF attacks while monitoring drug safety.

The significance of the study includes short and long-term benefits. Fewer FMF attacks will result in less functional impairment and a higher quality of life in colchicine resistant or intolerant patients. Once weekly injections have the potential to improve treatment compliance. Fewer acute attacks of arthritis may prevent the development of chronic joint damage. In the long-term, better FMF control may prevent amyloidosis. This study may confirm the importance of IL-1 in the pathogenesis of FMF and provide support for an FDA filing for use of Rilonacept in FMF. The study design may serve as a template for trials of new biologic drugs for rare diseases.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a definitive diagnosis of FMF as by the Tel-Hashomer clinical criteria (long version of criteria) with at least one mutation on one of the MEFV gene alleles. However, subjects with an isolated heterozygous mutation of exon 2 of the MEFV gene (including E148Q) will not be eligible.
* Subject must have an estimated mean of at least one acute FMF attack per month before and during the month of screening.
* Subject is at least four years of age (with no upper limit of age).
* Subjects must have received an adequate trial of colchicine defined as treatment of at least 1.5 mg/d for at least 3 months if ≥6 years old or 1.2 mg/d if less than 6 years, or an inability to tolerate colchicine due to adverse effects in a dose that controls acute attacks in the frequency of less than one attack per month.
* If subject is being treated with anakinra at the time of consent, washout must be done (about 3 days). Subject must experience 2 attacks before randomization visit can occur.
* If subject has been treated previously with anti-TNF drugs, appropriate washout must be done. Etanercept must be discontinued for 4 weeks prior to randomization; Adalimumab and Infliximab must be discontinued for 8 weeks prior to randomization.
* If subject is a female of childbearing potential, she must agree to use adequate contraception (adequate contraception can include abstinence) for the duration of the trial and 3 months after and must have a negative serum or urine pregnancy test prior to administration of study medication.
* If subject is a male and has reached puberty, he must agree to use adequate contraception or abstinence during the study and for 3 months after discontinuation from study.
* Subject's parent or legal guardian has provided written informed consent prior to screening for this study or if subject is older than 18 years has provided informed consent him/herself.
* Subject, if applicable, has assented to participate prior to screening for this study.
* Subject and, if applicable, parent/legal guardian, agree to comply with study requirements and are able to come to the clinic for all required study visits.

Exclusion Criteria:

* The subject has existing biopsy proven amyloidosis or proteinuria >0.5 gram per day.
* The subject has another active inflammatory rheumatic disease.
* The subject has an active malignancy of any type, or history of a malignancy.
* The subject has active GI disease (e.g., inflammatory bowel disease), a chronic or acute renal or hepatic disorder, or a significant coagulation defect.
* The subject has an AST (SGOT), ALT (SGPT) or BUN >2 x ULN or creatinine >1.5 mg/dL or any other laboratory abnormality considered by the examining physician to be clinically significant within 28 days before the Baseline visit.
* Current use of an anti-tumor necrosis factor drug.
* The subject has, in the investigator's opinion, a chronic condition (e.g., diabetes, epilepsy) that is either not stable or well-controlled and may interfere with the conduct of the study.
* The subject has received any investigational medication within 30 days before the first dose of study medication or is scheduled to receive an investigational drug, other than study medications described in this protocol, during the course of the study.
* The subject has chronic or active infection or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 30 days or oral antibiotics within 14 days prior to the screening evaluation.
* The subject has known positive human immunodeficiency virus (HIV) status.
* The subject has known past or current hepatitis.
* The subject has received a live virus vaccine within 1 month prior to the baseline visit.
* The subject has a positive PPD test.
* The subject is sexually active and not practicing effective birth control.
* The subject is pregnant or breast feeding a child.
* Any concurrent medical condition which would, in the investigator's opinion, compromise the subject's ability to tolerate the study drug or would make the subject unable to cooperate with the protocol.
* History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or give informed consent.
* Subject has a history of alcohol or drug abuse within the past 6 months that would interfere with ability to comply with protocol requirements.
* Inability to comply with the study requirements for any reason.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Hashkes, MD, MSc, Study Director — Shaare Zedek Medical Center/The Cleveland Clinic Foundation
Locations (5):
- United States (5):
  - Children's Hospital Los Angeles/Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Central California, Madera, California
  - NIH, Bethesda, Maryland
  - NYU Hospital for Joint Diseases, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Result] Hashkes PJ, Spalding SJ, Giannini EH, Huang B, Johnson A, Park G, Barron KS, Weisman MH, Pashinian N, Reiff AO, Samuels J, Wright DA, Kastner DL, Lovell DJ. Rilonacept for colchicine-resistant or -intolerant familial Mediterranean fever: a randomized trial. Ann Intern Med. 2012 Oct 16;157(8):533-41. doi: 10.7326/0003-4819-157-8-201210160-00003. PMID 23070486
- [Derived] Hashkes PJ, Spalding SJ, Hajj-Ali R, Giannini EH, Johnson A, Barron KS, Weisman MH, Pashinian N, Reiff AO, Samuels J, Wright D, Lovell DJ, Huang B. The effect of rilonacept versus placebo on health-related quality of life in patients with poorly controlled familial Mediterranean fever. Biomed Res Int. 2014;2014:854842. doi: 10.1155/2014/854842. Epub 2014 May 15. PMID 25147819
- [Derived] Huang B, Giannini EH, Lovell DJ, Ding L, Liu Y, Hashkes PJ. Enhancing crossover trial design for rare diseases: limiting ineffective exposure and increasing study power by enabling patient choice to escape early. Contemp Clin Trials. 2014 Jul;38(2):204-12. doi: 10.1016/j.cct.2014.05.001. Epub 2014 May 12. PMID 24833067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from October 2008 until February 2010. The study was conducted in 6 clinics in the United States in FMF clinics or clinics in regions where a higher prevalence of FMF is expected based on local population ethnicity.
Pre-assignment Details: Participants had an estimated mean ≥1 FMF attack/month for 3 months before screening, and ≥1 attack/month during screening/run-in period. There was a wash-out period of other biologic medications for those using them at screening. 2 subjects withdrew consent, one lacked mutations and one had insufficient attacks and were excluded before baseline.
Groups:
- Rilonacept-Placebo-Rilonacept-Placebo; Rilonacept-Placebo-Placebo-Rilonacept: Patients received in the randomized sequence above two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine. Overall study was 12 months.
- Placebo-Rilonacept-Placebo-Rilonacept; Placebo-Rilonacept-Rilonacept-Placebo: Patients received in the randomized sequence above two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine.
Period: 1st Course
Arm/Group | Rilonacept-Placebo-Rilonacept-Placebo | Rilonacept-Placebo-Placebo-Rilonacept | Placebo-Rilonacept-Placebo-Rilonacept | Placebo-Rilonacept-Rilonacept-Placebo
Started | 4 | 3 | 3 | 4
Completed | 3 (1 left after 1st course (transportation issues)) | 3 | 3 | 3 (Patient lost to follow-up towards end of 1st course)
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Period: 2nd Course
Arm/Group | Rilonacept-Placebo-Rilonacept-Placebo | Rilonacept-Placebo-Placebo-Rilonacept | Placebo-Rilonacept-Placebo-Rilonacept | Placebo-Rilonacept-Rilonacept-Placebo
Started | 3 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Period: 3rd Course
Arm/Group | Rilonacept-Placebo-Rilonacept-Placebo | Rilonacept-Placebo-Placebo-Rilonacept | Placebo-Rilonacept-Placebo-Rilonacept | Placebo-Rilonacept-Rilonacept-Placebo
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: 4th Course
Arm/Group | Rilonacept-Placebo-Rilonacept-Placebo | Rilonacept-Placebo-Placebo-Rilonacept | Placebo-Rilonacept-Placebo-Rilonacept | Placebo-Rilonacept-Rilonacept-Placebo
Started | 2 | 3 | 3 | 3
Completed | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients Received Both Rilonacept and Placebo: Patients received in randomized sequences two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine.
  Patients were randomized to 4 treatment sequences:
  1. rilonacept- placebo-rilonacept-placebo; 2. placebo-rilonacept-placebo-rilonacept 3. rilonacept- placebo-placebo-rilonacept and 4. placebo-rilonacept-rilonacept-placebo.
  Overall length of study for each participant is 12 months.
Arm/Group | All Patients Received Both Rilonacept and Placebo
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of Rilonacept in Decreasing the Number of Acute FMF Attacks.
Description: Difference in number of attacks per treatment month between rilonacept and placebo
Time Frame: attacks were assessed at the end of each 3 month treatment course (overall up to 6 month of rilonacept and 6 months of placebo, each)
Population: Patients who received at least one complete treatment course and reported attacks were analyzed for the primary outcome measure.
Measure: Median (Inter-Quartile Range); unit: number of attacks per month
Groups:
- Rilonacept; Placebo: Patients received in randomized sequences two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine.
  Patients were randomized to 4 treatment sequences:
  1. rilonacept- placebo-rilonacept-placebo; 2. placebo-rilonacept-placebo-rilonacept 3. rilonacept- placebo-placebo-rilonacept and 4. placebo-rilonacept-rilonacept-placebo.
  Overall length of study for each participant is 12 months.
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 12
number of attacks per month | 0.77 [0.18 to 1.20] | 2.00 [0.90 to 2.40]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Based upon FMF colchicine controlled studies showing an ~80% decrease in attacks, we estimated, based on baseline attacks every 4 weeks, there would be a difference of 0.5 attacks per month between rilonacept and placebo. With a two-sided 5% significance level and power of 80% we aimed for 14 evaluable participants who completed at least 2 treatment courses. The null hypothesis is that there would be no significant differences in the number of attacks between use of rilonacept and placebo; Test type: Superiority or Other; p = 0.027, Signed rank; Risk Ratio, log = -1.7, 95% CI 2-sided [-3.4 to -0.1], Standard Deviation 0.78
Statistical Analysis 2: Comparison: Rilonacept vs Placebo; This analysis was done by Bayesian Statistics using a non-informative (neutral) prior (log normal distribution mean 9 [SD 10]). The null hypothesis was that the rilonacept/placebo FMF odds ratio of attacks was 1; Test type: Superiority or Other; Bayesian modeling; Odds Ratio (OR) = 0.59, 95% CI [0.39 to 0.85], Standard Deviation 0.12 — Attacks while receiving rilonacept is the numerator and attacks while receiving placebo is the denominator. In Bayesian statistics credible interval equals confidence interval

2. Primary Outcome: To Determine if There is a Medically Important Difference Between the Safety Profiles of Rilonacept vs. Placebo.
Description: Differences in adverse events (AEs) between rilonacept and placebo per patient-month of treatment. We separately analyzed injection site reactions and infectious adverse events. Other adverse events were too small in number to analyze. The upper table (and first statistical analysis) regards injection site reactions and lower table (and second statistical analysis) regards infections.
Time Frame: 12 months of entire study length
Population: Safety analysis included all participants who received at least one dose of medication.
Measure: Median (Inter-Quartile Range); unit: AEs per patient-month of treatment
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 14
AEs per patient-month of treatment
  Injection site reactions | 1 [0 to 1.04] | 0 [0 to 0.36]
  Infections | 0 [0 to 0.12] | 0.18 [0 to 0.29]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There were no significant differences between rilonacept and placebo in the occurence of injection site reactions. No power calculations for this outcome; Test type: Superiority or Other; p = 0.047, Signed rank; Median Difference (Net) = 0, 95% CI 2-sided [-4 to 0], Standard Deviation 1.26
Statistical Analysis 2: Comparison: Rilonacept vs Placebo; Null hypothesis: There were no significant differences between rilonacept and placebo in the occurence of infections. No power calculations for this outcome; Test type: Superiority or Other; p = 0.13, Signed rank; Median Difference (Net) = 0, 95% CI 2-sided [-0.56 to 0.17]

3. Secondary Outcome: To Determine the Difference in the Length of Attacks During Treatment With Rilonacept vs. Placebo.
Description: This outcome was the difference in days in the length of attacks between rilonacept and placebo.
Time Frame: 12 months
Population: Participants who received any treatment and had recorded attacks
Measure: Median (95% Confidence Interval); unit: Number of days
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 14
Number of days | 2.8 [1 to 3.3] | 3.2 [2.7 to 4]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There were no significant differences in the length of attacks during rilonacept vs. placebo treatment courses. Since this was a secondary outcome there were no power calculations performed; Test type: Superiority or Other; p = 0.32, Signed rank; Mean Difference (Net) = -1.2, 95% CI [-2.4 to 0.5], Standard Deviation 0.5

4. Secondary Outcome: Percentage of Treatment Courses Without FMF Attacks in Rilonacept Courses as Compared to Placebo Courses.
Description: The percentage of rilonacept and placebo treatment courses without FMF attacks.
Time Frame: Each treatment course of up to 3 months
Population: Participants who at least one complete treatment course.
Measure: Number; unit: Percentage of courses
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of courses | 29 | 0
Statistical Analysis 1: Comparison: Rilonacept; Null hypothesis: There are no significant differences in the number of treatment courses without attacks between rilonacept and placebo. As a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.004, McNemar; Differences in percent of courses = 29

5. Secondary Outcome: To Determine the Proportion of Courses in Which Subjects Attained at Least a 50% Decrease in Acute FMF Attacks During Rilonacept Courses as Compared to Placebo Courses.
Description: Differences between rilonacept and placebo in the percentage of courses that attained at least a 50% decrease in FMF attacks when compared to attacks in the screening period.
Time Frame: Up to 3 months for each treatment course
Population: Participants who completed at least one complete treatment course.
Measure: Number; unit: Percentage of courses
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 13
Percentage of courses | 75 | 35
Statistical Analysis 1: Comparison: Rilonacept; Null hypothesis: There are no significant differences in the number of treatment courses attaining at least a 50% decrease in attacks when compared to baseline between rilonacept and placebo courses.Since this was a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.006, McNemar; Difference in percent of courses = 40

6. Secondary Outcome: To Determine Differences in the Time to the Development of Attacks Between the Treatment Arms (Rilonacept vs. Placebo).
Description: In a survival analysis we measured the difference (in days) until the development of the first and second attack within a treatment course of up to 3 months and examined differences in this parameter between rilonacept and placebo. Data regarding the development of the second attack are reported below. In regards to the first attack there were no significant differences between rilonacept and placebo (20 days (7.5,>90)for rilonacept; 15 (8,32) for placebo, P=0.066).
Time Frame: 3 months
Population: All participants who received an intervention and developed an attack were analyzed.
Measure: Median (Inter-Quartile Range); unit: days until second attack
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 13 | 14
days until second attack | 90 [25 to 90] | 36 [15 to 68]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There were no significant differences between rilonacept and placebo in the number of days from the start of the treatment course until the development of the a second attack; Test type: Superiority or Other; p = 0.009, Kaplan-Meier survival analysis; Log Rank = 0.009

7. Secondary Outcome: To Determine the Differences in the Erythrocyte Sedimentation Rate Between the Treatment Arms (Rilonacept vs. Placebo).
Description: Erythrocyte sedimentation rate - ESR (mm/h)
Time Frame: 3 months (each treatment course, overall 12 months)
Population: Participants who completed at least one treatment course of both rilonacept and placebo.
Measure: Median (Inter-Quartile Range); unit: mm/h
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
mm/h | 5.8 [2 to 16] | 14 [7 to 19]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no significant differences in the erythrocyte sedimentation rate between rilonacept and placebo. As a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.156, Signed Rank; Median Difference (Net) = 6.5, 95% CI 2-sided [-0.5 to 12.5]

8. Secondary Outcome: To Determine the Differences in C-Reactive Protein Between the Treatment Arms (Rilonacept vs. Placebo)
Description: Differences between the treatment courses in the C-Reactive Protein levels mg/L
Time Frame: 3 months (each treatment course, overall 12 months)
Population: Patients who received at least one course each of rilonacept and placebo
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
mg/L | 2 [2 to 4] | 4 [2 to 9]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no differences in the C-reactive protein levels between the treatment courses. Since this was a secondary outcome measure no power calculations were performed; Test type: Superiority or Other; p = 0.22, Signed Rank; Median Difference (Net) = 0.04, 95% CI 2-sided [-0.03 to 0.29]

9. Secondary Outcome: To Determine the Differences in the Platelet Count Between the Treatment Arms (Rilonacept vs. Placebo)
Description: The difference between the treatment arms in the platelet count X 10 to the power of 9
Time Frame: 3 months (each treatment course, overall 12 months)
Population: The number of patients who received at least one course each of rilonacept and placebo
Measure: Median (Inter-Quartile Range); unit: cell count X10 to the power of 9
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
cell count X10 to the power of 9 | 262 [246 to 318] | 334 [305 to 352]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There were no differences between the platelet count between the rilonacept and placebo courses. Since this was a secondary outcome no power calculations were performed; Test type: Superiority or Other; p = 0.078, Signed Rank; Median Difference (Net) = 29.4, 95% CI 2-sided [0.4 to 78.1]

10. Secondary Outcome: To Determine the Differences in the Fibrinogen Levels Between the Treatment Arms (Rilonacept vs. Placebo)
Description: The differences between treatment arms in the fibrinogen level (micromol/L)
Time Frame: 3 months (each treatment course, overall 12 months)
Population: Patients who received at least one course each of rilonacept and placebo
Measure: Median (Inter-Quartile Range); unit: micromol/L
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
micromol/L | 6.56 [6.41 to 9.70] | 9.56 [9.26 to 10.17]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no differences between the treatment arms in the fibrinogen level. Since this was a secondary outcome no power calculations were performed; Test type: Superiority or Other; p = 0.063, Signed Rank; Median Difference (Net) = 108, 95% CI 2-sided [6.5 to 139.5]

11. Secondary Outcome: To Determine the Differences in Serum Amyloid A Levels Between the Treatment Arms (Rilonacept vs. Placebo)
Description: The difference between the treatment arms in serum amyloid A levels (mg/L)
Time Frame: 3 months (each treatment course, overall 12 months)
Population: Patients who received at least one course each of rilonacept and placebo
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
mg/L | 13 [0 to 40] | 15 [0 to 192]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no differences between the treatment arms in the serum amyloid A levels. Since this was a secondary outcome no power calculations were performed; Test type: Superiority or Other; p = 0.50, Signed Rank; Median Difference (Net) = 0, 95% CI 2-sided [-4 to 0]

12. Secondary Outcome: To Determine the Differences in the Quality of Life Between the Treatment Arms (Rilonacept vs. Placebo).
Description: Differences in the health-related quality of life (HRQOL) during treatment with rilonacept vs. placebo. HRQOl was measured by the Childhood Health Questionnaire which was adopted also for adults. There are 2 summary scores: 1. Physical summary score. 2. Psychosocial summary score. The data reported below in the upper table is the physical summary composite score and in the lower table the psychosocial summary composite score. Scores were from 0-100 (higher is better) with a score of 50 representing the mean of the normal population.
Time Frame: 12 months
Population: Participants who received at least one treatment course of rilonacept and placebo.
Measure: Median (Inter-Quartile Range); unit: Composite HRQOL summary score
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
Composite HRQOL summary score
  Physical HRQOL summary composite score | 33 [25.8 to 38.1] | 20.3 [10.5 to 32.7]
  Psychosocial HRQOL summary composite score | 53.3 [48.6 to 57.2] | 49.8 [42.5 to 59]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no significant differences in the physical health-related quality of life between rilonacept and placebo. As a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.021, Signed rank; Median Difference (Net) = -6.5, 95% CI 2-sided [-11.1 to -2.3]
Statistical Analysis 2: Comparison: Rilonacept vs Placebo; Test type: Superiority or Other; p = 0.42, Signed Rank; Median Difference (Net) = -4.2, 95% CI 2-sided [-6.8 to 3.9]

13. Secondary Outcome: To Determine the Differences in the FMF Severity Score of the Subjects Between the Treatment Arms (Rilonacept vs. Placebo).
Description: Differences in the Armenian Evaluation Score between rilonacept and placebo courses. The Armenian Evaluation Score is a composite score of disease severity based on the frequency, duration and character of attacks (degree of fever and severity of serositis). It was adapted to calculate a score for a 3-month treatment course. The lowest (best) score is 0 and higher values are worse. In theory there is no upper limit to the scale. The total score is reported (there are no subscales).
Time Frame: overall 12 months
Population: Participants who received at least one course each of placebo and rilonacept.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 5.5 [3 to 13] | 11 [7.8 to 12.5]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no significant differences in the FMF Armenian Evaluation (severity) Score between rilonacept and placebo. As a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.136, Signed rank; Median Difference (Net) = 2.5, 95% CI 2-sided [-2.3 to 9.8]

14. Secondary Outcome: To Determine the Differences in the Proportion of Time Subjects Received Rilonacept vs Placebo
Description: The proportion of time within the trial that participants received rilonacept as opposed to placebo. The reason for this outcome is that participants who had at least 2 attacks within an individual treatment course were able to "escape" in a blinded manner to the other treatment arm until the end of that treatment course and then resume the original randomization sequence. Thus participants may have been treated for a longer time with one treatment arm or the other.
Time Frame: 12 months
Population: Participants who received at least one treatment course of both rilonacept and placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of time treated
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 12 | 12
Percentage of time treated | 52.5 [50.5 to 70.5] | 47.5 [29.5 to 49.5]
Statistical Analysis 1: Comparison: Rilonacept vs Placebo; Null hypothesis: There are no significant differences in the proportion of time participants were treated with rilonacept and placebo. As a secondary measure there were no power calculations; Test type: Superiority or Other; p = 0.089, Signed rank; Median Difference (Net) = -5, 95% CI 2-sided [-15 to -1]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Placebo: Adverse events during placebo treatment. Patients received in randomized sequences two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine.
  Patients were randomized to 4 treatment sequences:
  1. rilonacept- placebo-rilonacept-placebo; 2. placebo-rilonacept-placebo-rilonacept 3. rilonacept- placebo-placebo-rilonacept and 4. placebo-rilonacept-rilonacept-placebo.
- Rilonacept: Adverse events during rilonacept treatment. Patients received in randomized sequences two 3-month courses of rilonacept (IL-1 Trap),2.2 mg/kg/wk (max 160 mg) by SC injection and two 3-month courses of equal volume placebo by weekly SC injection. This was in addition to the pre-study dose of colchicine.
  Patients were randomized to 4 treatment sequences:
  1. rilonacept- placebo-rilonacept-placebo; 2. placebo-rilonacept-placebo-rilonacept 3. rilonacept- placebo-placebo-rilonacept and 4. placebo-rilonacept-rilonacept-placebo.
Arm/Group | Placebo | Rilonacept
Serious Adverse Events (participants affected / at risk) | 3/14 | 3/13
Other Adverse Events (participants affected / at risk) | 12/14 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Rilonacept (N=13)
Hospitalization for FMF attack (Immune system disorders) | 2 (3) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Rilonacept (N=13)
Injection site reaction (Injury, poisoning and procedural complications) | 5 (13) | 7 (53)
Upper respiratory infection/Otitis (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes labialis (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Epstein Barr virus (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (General disorders) | 0 (0) | 1 (2)
Headaches (Nervous system disorders) | 1 (1) | 1 (1)
Otitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia/bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (3)
Asthma attack (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea, vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Heat and cold sensitivity (General disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Fracture - toe (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Facial edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sore throat (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Alanine aminotransferase (ALT) elevation (Investigations) | 0 (0) | 1 (1)
Creatine Kinase (CPK) elevation (Investigations) | 1 (1) | 0 (0)
Overactive bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Facial skin infection (Infections and infestations) | 1 (1) | 0 (0)
Nose bleed (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Oral thrush (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Small sample size - accounted for in study design and analysis plan.
2. Carry over/lag effect of rilonacept - sensitivity analysis of shifting course time frame showed similar results.
3. Heterogeneity of FMF mutations
4. Different age groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No